CLINICAL TRIAL: NCT01696422
Title: Phase II, Step-wise, Randomized, Double-blind, Controlled Clinical Trial for Safety and Immunogenicity Evaluation of a Lyophilized Formulation of Dengue 1,2,3,4 (Attenuated) Vaccine in Healthy Adults
Brief Title: Phase II Trial to Evaluate Safety and Immunogenicity of a Dengue 1,2,3,4 (Attenuated) Vaccine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Butantan Institute (Other Government)
Collaborators: Banco Nacional de Desenvolvimento Economico e Social (Unknown); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Butantan Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DEN-01-IB; U1111-1135-4553 (Registry Identifier: UTN)
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Dengue
Keywords: Dengue; tetravalent attenuated Vaccine; Healthy adults
MeSH Terms: conditions — Dengue | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Step A: dengue lyophilized vaccine (Experimental): Dengue 1,2,3,4 (attenuated) vaccine Two doses with a six-months interval, SC
  Interventions: Biological: Dengue 1,2,3,4 (attenuated) vaccine
- Step A:dengue liquid vaccine (Active Comparator): TetraVax-DV Vaccine - Admixture TV003 Two doses with a six-months interval, SC
  Interventions: Biological: TetraVax-DV Vaccine - Admixture TV003
- Step A: Placebo (Placebo Comparator): Placebo comparator Two doses with a six-months interval, SC
  Interventions: Other: Placebo
- Step B: dengue lyophilized vaccine (Experimental): Dengue 1,2,3,4 (attenuated) vaccine Single dose, SC
  Interventions: Biological: Dengue 1,2,3,4 (attenuated) vaccine
- Step B: Placebo (Placebo Comparator): Placebo comparator Single dose, SC
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Dengue 1,2,3,4 (attenuated) vaccine — Dose 1000 PFU per virus (1,2,3,4) Route:subcutaneous
  Other Names: Butantan DV; Dengue Tetravalent Vaccine - Lyophilized formulation
  Arms: Step A: dengue lyophilized vaccine; Step B: dengue lyophilized vaccine
Biological: TetraVax-DV Vaccine - Admixture TV003 — Dose 1000 PFU per virus (1,2,3,4) Route: subcutaneous
  Other Names: Dengue Tetravalent Vaccine - Liquid formulation
  Arms: Step A:dengue liquid vaccine
Other: Placebo — Route:subcutaneous
  Arms: Step A: Placebo; Step B: Placebo

SUMMARY:
This is a phase II step-wise, randomized, multicenter, double-blind and controlled clinical trial to evaluate the safety and immunogenicity of a attenuated tetravalent lyophilized dengue vaccine manufactured by Butantan Institute. Three Clinical Sites at University of Sao Paulo - Brazil will participate in the study. A total of 300 volunteers will be recruited and divided into two steps: Step A (with no previous exposure to dengue) and Step B (with and without previous exposure to dengue). In step A the participants will be assigned to receive either the lyophilized vaccine, or the liquid vaccine(developed at NIH and produced and formulated at Butantan according to the NIH-Protocol), or the placebo. In Step B participants will be assigned to receive either the lyophilized vaccine, or the placebo. Both vaccine formulations (lyophilized and liquid) are composed of the same attenuated viruses: rDEN1∆30, rDEN2/4∆30(ME), rDEN3∆30/31, and rDEN4∆30. At the end of the study, 20 volunteers will have received the liquid formulation (NIH), 210 the lyophilized formulation (Butantan), and 70 will have received the placebo. All participants included in both steps will be followed by a period of five years after their inclusion in the study. The study hypothesis is that the investigational lyophilized dengue vaccine manufactured by Butantan Institute is safe and confers balanced immune response, after one dose of 1000PFU, to all for vaccine viruses.

DETAILED DESCRIPTION:
This is a phase II step-wise, randomized, multicenter, double-blind and controlled clinical trial to evaluate the safety and immunogenicity of an attenuated tetravalent lyophilized dengue vaccine manufactured by Butantan Institute. A total of 300 volunteers will be recruited including men and no pregnant/breastfeeding women between 18 and 59 years of age complete, with and without previous exposure to dengue that will be randomized into Step A and Step B. Step A will include 50 volunteers with no previous exposure and they will be randomly assigned to receive one dose of either the lyophilized formulation (Butantan), or the liquid formulation (TetraVax-DV Vaccine - Admixture TV003 developed by NIH/NIAID and produced and formulated at Butantan according the NIH-Protocol), or the placebo. A second dose will be administered six months after the first vaccination as part of an exploratory assessment. Step B will include 250 participants(50 without previous exposure to dengue,and 200 with previous exposure to dengue) who will be randomly assigned to receive one dose of either the lyophilized formulation (Butantan),or the placebo. All participants included in both steps will be followed by a period of five years after their inclusion in the study. The vaccines will be administered at dose of 1000 PFU (for each of the vaccine viruses),and both vaccines and the placebo will be administered subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (men and non-pregnant women), from 18 to 59 years old;
* Willingness to participate throughout the study period (approximately five years);
* Willingness to participate documented by the signature of ICF;
* Females with childbearing potential must be willing to avoid pregnancies up to three weeks after the last vaccine dose. All female volunteers will be considered with childbearing potential unless they have documented history of hysterectomy, tubal ligation or are postmenopausal (12 months of amenorrhea after the last menstrual period).

Exclusion Criteria:

* Pregnancy (confirmed by positive beta-hCG test) or breastfeeding;
* Evidence of active neurological, cardiac, pulmonary, hepatic or renal disease as clinical history, physical examination and/or laboratory results;
* Compromised immune system diseases including: diabetes mellitus, cancer (except basal cell carcinoma) and autoimmune diseases;
* Behavioral, cognitive or psychiatric disease that in the opinion of the principal investigator or his representative physician, affects the participant ability to understand and cooperate with all study protocol requirements;
* Values of absolute neutrophil, alanine aminotransferase (ALT) or serum creatinine count greater than or equal to Grade 1, as defined in the protocol;
* Abusive usage of alcohol or drugs in the past 12 months that has caused medical, professional or family problems, indicated by clinical history;
* History of severe allergic reactions or anaphylaxis;
* Diagnosis of asthma with a history of hospitalization in the last six months due to illness;
* Fever or suspect fever within 72 hours prior to vaccination or axillary temperature greater than 37,8°C on the day of vaccination;
* Positive result of HIV-1 serology by screening or confirmed tests;
* Screening or confirmed positive test for hepatitis C virus (HCV);
* Positive test of hepatitis B virus antigen surface (AgHBs) alone or against hepatitis B "core" antigen antibody (anti-HBc);
* Use of corticosteroids (except topical or nasal) or other immunosuppressive drugs within 42 days before study initiation/baseline. It will be considered immunosuppressive dose of corticosteroids the equivalent to a dose ≥10 mg of prednisone per day for over 14 days;
* Use of anticoagulant medication;
* Have received live virus vaccine within 28 days or killed virus vaccine in the last 14 days prior to vaccination, or have a scheduled immunization during the first 42 days after receiving the investigational product;
* History of asplenia;
* Have received blood products in the past six months, including transfusions or immunoglobulin, or scheduled administration of blood products or immunoglobulin for the first 42 days after vaccination;
* Use of any investigational product within 42 days before or after receiving this study vaccination;
* Has participated in another clinical trial six months prior to vaccination;
* Denies permission for biological material storage for future research as defined in ICF;
* Any other condition that might put in risk the safety/rights of a potential participant or hurdle his/her compliance with this protocol in investigator's opinion or his representative physician.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Safety | Up to day 21 after vaccination
  Frequency of solicited and unsolicited local and systemic adverse reactions up to Day 21 after vaccination.
Immunogenicity | Up to day 91 after vaccination
  Seroconversion rate for each of the four vaccine viruses defined by PRNT50 ≥1:10 for each vaccine virus serotype on Days 28, 56 or 91.

SECONDARY OUTCOMES:
Safety | up to Day 182 after the first vaccination
  1. Unsolicited adverse events after Day 21 and up to Day 182 after the first vaccination;
  2. Viremia for each of the four vaccine virus on Days 3, 6, 9, 12, 15 and 21 after the first vaccination of all volunteers in Step A of study and 40 volunteers with previous exposure to Dengue of Step B. For other volunteers from Step B, viremia only is measured on Day 12.
  3. Cases of suspected and confirmed dengue in five years after the first vaccination;
Immunogenicity | Annualy up to five years
  1. Response rates of monovalent, bivalent, trivalent or tetravalent, at Day 28, 56 and 91 and annually after vaccination, as measured by PRNT50 for each one of the four vaccine viruses;
  2. The difference between the geometric means, pre and post vaccination, serum level of neutralizing antibodies measured by PRNT50 for each of the four vaccine viruses evaluated until five years after the first vaccination.

OTHER OUTCOMES:
Exploratory | Up to Day 182 after the second vaccination
  1. The seroconversion rate for each one of the four vaccine according to previous exposure to other flaviviruses;
  2. The solicited and unsolicited local and systemic adverse reactions, until Day 21 after the second vaccination;
  3. Unsolicited adverse events after Day 21 and Day 182 after the second vaccination for participants from Step A;
  4. The differences in pre and post vaccination cellular immune response after the first and second vaccination and annually for five years for participants in Step A;
  5. Viremia for each one of the four vaccine viruses on Days 3, 6, 9, 12, 15 and 21 after a second vaccination for participants in Step A;
  6. The difference in rates of seroconversion for each of the four types vaccination after the second vaccination for participants in Step A;
  7. The differences in cellular immune response pre and post vaccination after the first vaccination and annually for five years for 40 participants from Step B with previous exposure to dengue.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander R Precioso, MD, PhD, Study Director — Instituto Butantan
Locations (2):
- Brazil (2):
  - Instituto da Criança do Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo

REFERENCES:
- [Background] Blaney JE Jr, Durbin AP, Murphy BR, Whitehead SS. Development of a live attenuated dengue virus vaccine using reverse genetics. Viral Immunol. 2006 Spring;19(1):10-32. doi: 10.1089/vim.2006.19.10. PMID 16553547
- [Background] Durbin AP, Kirkpatrick BD, Pierce KK, Schmidt AC, Whitehead SS. Development and clinical evaluation of multiple investigational monovalent DENV vaccines to identify components for inclusion in a live attenuated tetravalent DENV vaccine. Vaccine. 2011 Sep 23;29(42):7242-50. doi: 10.1016/j.vaccine.2011.07.023. Epub 2011 Jul 21. PMID 21781997
- [Background] Durbin AP, Kirkpatrick BD, Pierce KK, Elwood D, Larsson CJ, Lindow JC, Tibery C, Sabundayo BP, Shaffer D, Talaat KR, Hynes NA, Wanionek K, Carmolli MP, Luke CJ, Murphy BR, Subbarao K, Whitehead SS. A single dose of any of four different live attenuated tetravalent dengue vaccines is safe and immunogenic in flavivirus-naive adults: a randomized, double-blind clinical trial. J Infect Dis. 2013 Mar 15;207(6):957-65. doi: 10.1093/infdis/jis936. Epub 2013 Jan 17. PMID 23329850
- [Derived] Silveira CGT, Magnani DM, Costa PR, Avelino-Silva VI, Ricciardi MJ, Timenetsky MDCST, Goulart R, Correia CA, Marmorato MP, Ferrari L, Nakagawa ZB, Tomiyama C, Tomiyama H, Kalil J, Palacios R, Precioso AR, Watkins DI, Kallas EG. Plasmablast Expansion Following the Tetravalent, Live-Attenuated Dengue Vaccine Butantan-DV in DENV-Naive and DENV-Exposed Individuals in a Brazilian Cohort. Front Immunol. 2022 Jun 28;13:908398. doi: 10.3389/fimmu.2022.908398. eCollection 2022. PMID 35837409
- [Derived] Kallas EG, Precioso AR, Palacios R, Thome B, Braga PE, Vanni T, Campos LMA, Ferrari L, Mondini G, da Graca Salomao M, da Silva A, Espinola HM, do Prado Santos J, Santos CLS, Timenetsky MDCST, Miraglia JL, Gallina NMF, Weiskopf D, Sette A, Goulart R, Salles RT, Maestri A, Sallum AME, Farhat SCL, Sakita NK, Ferreira JCOA, Silveira CGT, Costa PR, Raw I, Whitehead SS, Durbin AP, Kalil J. Safety and immunogenicity of the tetravalent, live-attenuated dengue vaccine Butantan-DV in adults in Brazil: a two-step, double-blind, randomised placebo-controlled phase 2 trial. Lancet Infect Dis. 2020 Jul;20(7):839-850. doi: 10.1016/S1473-3099(20)30023-2. Epub 2020 Mar 24. PMID 32220283